CLINICAL TRIAL: NCT04141605
Title: Global Utilization and Registry Database for Improved Heart Preservation
Acronym: GUARDIAN
Status: Enrolling by invitation | Type: Observational
Sponsor: Paragonix Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: PGX-002
Record Dates: First submitted 2019-10-16; First posted 2019-10-28 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Heart Diseases; Heart Failure; Heart Defects, Congenital
MeSH Terms: conditions — Heart Diseases; Heart Failure; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- SherpaPak CTS Patients: Patients whose donor heart was transported with the SherpaPak CTS
  Interventions: Device: SherpaPak Cardiac Transport System
- Standard Transport Patients: Patients whose donor heart was transported with a method other than SherpaPak CTS in the past two years

INTERVENTIONS:
Device: SherpaPak Cardiac Transport System — The Paragonix SherpaPak Cardiac Transport System ("SherpaPak CTS") is an ultraportable hypothermic preservation and transport system intended for use with donor hearts. The device is a legally marketed, FDA cleared medical device in the United States and CE Marked medical device in the European Union.
  The SherpaPak CTS consists of multiple components: 1) outer transport shipper which contains within various non-ice based temperature controlled packaging elements, 2) an inner and outer hard shell assembly which provides a rigid barrier enclosure in which the heart is immersed and suspended in a cold storage solution cleared for use in storing and transporting donor hearts, 3) a data logger that monitors and displays the temperature of the cold storage solution in which the heart is stored during transport, and 4) four size heart connectors designed to accommodate various size aortic stem diameters by which donor hearts are attached.
  Other Names: SherpaPak CTS
  Groups: SherpaPak CTS Patients

SUMMARY:
The primary objective of this study is to collect real-world clinical performance data to assess the clinical outcomes of patients receiving heart transplants using donor hearts transported via the SherpaPak CTS System. These results will be compared to outcomes of retrospective patients whose hearts were transported with the previous standard method.

DETAILED DESCRIPTION:
This study is a registry study collecting data both retrospectively from patients already transplanted and prospectively from consecutively enrolled patients for heart transplantation. The study is a chart review study.

Ongoing eligible recipients will undergo heart transplantation according to standard practices at each participating institution.

This study will be conducted at an estimated 25 institutions globally and will have about up to 3000 patients. Subjects will be followed from transplant through one-year post-transplantation (i.e., 24 hours post-transplant, discharge, 30-days, 1-year, 2-years, 3-years, 4-years, 5-years).

GUARDIAN provides critical and contemporary data on patient outcomes, with additional insight into risk factors and patient-related indices. Both donor and recipient information along with procedural details (including transportation) will be collected to provide information for major discrete endpoints such as death, primary graft dysfunction, right ventricular dysfunction, CPB weaning, Inotrope use, CAV diagnosis, rejection, and survival.

Information about re-hospitalizations and re-transplantations is vital to address the integrated endpoint of days alive out of hospital, which is particularly relevant for this patient population. In addition, the number of in-hospital days and ICU time is closely tracked as the major resource utilized, after the initial transplant.

ELIGIBILITY:
Inclusion Criteria:

* Donor and donor hearts matched to the prospective recipient based upon institutional medical practice
* Registered male or female primary heart transplant candidates including pediatric candidates

Exclusion Criteria:

* Donor and donor hearts that do not meet institutional clinical requirements for transplantation
* When safe connection with the aorta cannot be made, e.g., due to lack of enough length of the aortic root
* Patients who are incarcerated persons (prisoners)
* Patients who have had a previous organ transplant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients registered on the heart transplant registry who receive a heart transplant at a participating center and do not meet any of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-02-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Primary Graft Dysfunction | one year
  Less than 40% LVEF by echocardiography or hemodynamics with RAP greater than 15 mm Hg, PCWP greater than 20 mm Hg, CI less thann 2 L/min/m^2, hypotension with MAP less than 70 mm Hg (lasting more than 1 hour)
Number of Patients with Right Ventricular Dysfunction | one year
  hemodynamics with RAP grater than 15mm Hg, PCWP less than 15 mm Hg, CI less than 2 L/min/m^2, TPG less than 15mm Hg/pulmonary artery systolic pressure less than 50 mmHg OR need for RVAD
Length of ICU Stay | one year
  Length of time patient admitted to the intensive care unit post transplant
Length of Hospital Stay | one year
  Length of time before patient is discharged from the hospital post transplant
Survival | 5 years
  The length of patient survival up to 5 years will be compared

SECONDARY OUTCOMES:
Hospitalizations | one year
  Number of related hospitalizations post transplant
CAV development | five years
  Number of patients who developed CAV between 1 and 5 years post transplant will be compared
Retransplant | five years
  The number of patients who were retransplanted will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Zuckermann, MD, Principal Investigator — ALLGEMEINES KRANKENHAUS WIEN
Locations (22):
- United States (17):
  - Stanford University, Stanford, California
  - Medstar Washington Hospital, Washington D.C., District of Columbia
  - University of Florida Health Shands Hospital, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Lutheran Hospital, Fort Wayne, Indiana
  - Kansas University Medical Center, Lawrence, Kansas
  - Tufts University Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Spectrum Health, Grand Rapids, Michigan
  - NewYork-Presbyterian Columbia University Irving Medical Center, New York, New York
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Pennslyvania State University, State College, Pennsylvania
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Sentara Healthcare, Norfolk, Virginia
- Austria (2):
  - University of Graz, Graz
  - Allgemeines Krankenhaus Wien, Vienna
- Spain (2):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clínico Universitario de Valladolid, Valladolid
- Manchester University, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will only be released as a summary of the results found at each center and overall. No individual patient data will be released.

REFERENCES:
- [Derived] Lerman JB, Patel CB, Casalinova S, Nicoara A, Holley CL, Leacche M, Silvestry S, Zuckermann A, D'Alessandro DA, Milano CA, Schroder JN, DeVore AD. Early Outcomes in Patients With LVAD Undergoing Heart Transplant via Use of the SherpaPak Cardiac Transport System. Circ Heart Fail. 2024 May;17(5):e010904. doi: 10.1161/CIRCHEARTFAILURE.123.010904. Epub 2024 Apr 11. PMID 38602105
- [Derived] D'Alessandro D, Schroder J, Meyer DM, Vidic A, Shudo Y, Silvestry S, Leacche M, Sciortino CM, Rodrigo ME, Pham SM, Copeland H, Jacobs JP, Kawabori M, Takeda K, Zuckermann A. Impact of controlled hypothermic preservation on outcomes following heart transplantation. J Heart Lung Transplant. 2024 Jul;43(7):1153-1161. doi: 10.1016/j.healun.2024.03.010. Epub 2024 Mar 19. PMID 38503386
- [Derived] Moayedifar R, Shudo Y, Kawabori M, Silvestry S, Schroder J, Meyer DM, Jacobs JP, D'Alessandro D, Zuckermann A. Recipient Outcomes With Extended Criteria Donors Using Advanced Heart Preservation: An Analysis of the GUARDIAN-Heart Registry. J Heart Lung Transplant. 2024 Apr;43(4):673-680. doi: 10.1016/j.healun.2023.12.013. Epub 2023 Dec 30. PMID 38163452
- [Derived] Shudo Y, Leacche M, Copeland H, Silvestry S, Pham SM, Molina E, Schroder JN, Sciortino CM, Jacobs JP, Kawabori M, Meyer DM, Zuckermann A, D'Alessandro DA. A Paradigm Shift in Heart Preservation: Improved Post-transplant Outcomes in Recipients of Donor Hearts Preserved With the SherpaPak System. ASAIO J. 2023 Nov 1;69(11):993-1000. doi: 10.1097/MAT.0000000000002036. Epub 2023 Apr 5. PMID 37678260